CLINICAL TRIAL: NCT03781401
Title: Blood Pressure Telemonitoring in Local Pharmacies and Blood Pressure Control in the Community
Brief Title: Telemonitoring of Blood Pressure in Local Pharmacies
Acronym: TEMPLAR
Status: Recruiting | Type: Observational
Sponsor: Italian Institute of Telemedicine (Other)
Collaborators: Italian Society of Hypertension (Other); Italian Society of General Practitioners (Unknown); Biotechmed Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: TEMPLAR
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring

SUMMARY:
The TEMPLAR project is an observational, cross-sectional, multicenter study involving several community pharmacies spread all over Italy. The aim of the project, the currently largest Italian ABPM Registry, is to analyze the 24-hour ABPMs performed in community pharmacies enabled for this service in accordance with the current Italian regulations, in order to evaluate the level of BP control in the community and to provide scientific evidence on the usefulness of a telehealth network involving the pharmacist for the screening and control of hypertension.

DETAILED DESCRIPTION:
The recent introduction of second-level services in Pharmacy, has resulted in the gradual diffusion of some techniques, which, under medical supervision, have enormous potential in improving screening, prevention and control of the most common chronic diseases. Among these services, 24-hour and home blood pressure monitoring are the most commonly available. The introduction of blood pressure monitoring in Pharmacy, under medical prescription, supervision and reporting, plays an important scientific role. As a matter of fact, the collected data can be useful for taking a picture of the status of the blood pressure control in a setting different from that of the Hospital or Hypertension Clinic. These data can also help to evaluate the usefulness of such a service in terms of improvement of public health and as a support to Doctor's intervention.

The aim of the project is to assess the level of blood pressure control in patients undergoing 24-hour or home blood pressure monitoring through Pharmacies enabled for this service in accordance with the current local laws. Specific objectives of the project are: a) to verify whether such a service is really useful in terms of hypertension screening, b) to assess the real blood pressure control of hypertensive patients pharmacologically treated, c) to typify the degree of blood pressure control according to the main demographic and clinical characteristics of the subjects.

This is an observational, cross-sectional, multicenter study involving Pharmacies spread all over Italy. These Pharmacies already make use of a telemonitoring and telereporting system based on 24-hour and home blood pressure monitoring, with centralized data collection. The service is developed in accordance with the rules governing the second-level services payable in Pharmacy (DL 03/10/2009 n. 153 and DM 16/12/2010) and with the legislation on protection of personal data (DL 30/06/2003 n. 196). The service is provided in accordance with the current Guidelines of the Italian Society of Hypertension and the European Society of Hypertension and is managed by Doctors expert of the methodology. The service is offered to patients upon payment and the test is prescribed by the General Practitioner (referring physician of the patient). The data collected as part of the service provided by the single Pharmacies are analyzed for the purposes of the Project. The project foresees the analysis of blood pressure recordings and clinical data of subjects of both sexes, aged ≥ 18 years, undergoing a 24-hour or home blood pressure monitoring because of a suspected hypertension (patients not pharmacologically treated) or to verify the degree of blood pressure control with antihypertensive drug therapy (patients under treatment).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients of both sexes and of any age
* Conventional clinical indications for ABPM (either treated with antihypertensive drugs or untreated)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients of both sexes and of any age with conventional clinical indications for ABPM (either treated with antihypertensive drugs or untreated) referred to the pharmacy by their family doctors for diagnostic purposes (established or suspected arterial hypertension).
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2010-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
24-hour blood pressure control rate | 10 years
  The percentage of patients with an average 24-hour blood pressure <130/80 mmHg

SECONDARY OUTCOMES:
Office blood pressure control rate | 10 years
  The percentage of patients with an office blood pressure <140/90 mmHg
Day-time blood pressure control rate | 10 years
  The percentage of patients with an average day-time blood pressure <135/85 mmHg
Night-time blood pressure control | 10 years
  The percentage of patients with an average night-time blood pressure <120/70 mmHg
Evaluation of blood pressure control in treated vs. untreated subjects | 10 years
  The percentage of treated vs. untreated patients with blood pressure control
Rate of patients with white-coat hypertension | 10 years
  Percentage of patients with an office SBP ≥140 mmHg and/or DBP ≥90 mmHg + 24-hour average BP <130/80 mmHg + day-time average BP <135/85 mmHg + night-time average BP <120/70 mmHg
Rate of patients with masked hypertension | 10 years
  Percentage of patients with an office BP <140/90 mmHg + 24-hour average SBP ≥130 mmHg and/or DBP ≥80 mmHg or day-time average SBP ≥135 mmHg and/or DBP ≥85 mmHg or night-time average SBP ≥120 mmHg and/or DBP ≥70 mmHg
Blood pressure control in subgroups at risk | 10 years
  Rate of office and ambulatory blood pressure control according to sex, age, cardiovascular risk factors and concomitant diseases

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Omboni, MD, Study Director — Italian Institute of Telemedicine
Locations (1):
- Italian Institute of Telemedicine, Solbiate Arno, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Omboni S, Mancinelli A, Rizzi F, Parati G; TEMPLAR (TEleMonitoring of blood Pressure in Local phARmacies) Project Group. Telemonitoring of 24-Hour Blood Pressure in Local Pharmacies and Blood Pressure Control in the Community: The Templar Project. Am J Hypertens. 2019 Jun 11;32(7):629-639. doi: 10.1093/ajh/hpz049. PMID 30976783
- [Result] Omboni S, Tenti M. Telepharmacy for the management of cardiovascular patients in the community. Trends Cardiovasc Med. 2019 Feb;29(2):109-117. doi: 10.1016/j.tcm.2018.07.002. Epub 2018 Jul 12. PMID 30037524
- [Result] Omboni S, Caserini M, Coronetti C. Telemedicine and M-Health in Hypertension Management: Technologies, Applications and Clinical Evidence. High Blood Press Cardiovasc Prev. 2016 Sep;23(3):187-96. doi: 10.1007/s40292-016-0143-6. Epub 2016 Apr 12. PMID 27072129
- [Result] Omboni S, Sala E. The pharmacist and the management of arterial hypertension: the role of blood pressure monitoring and telemonitoring. Expert Rev Cardiovasc Ther. 2015 Feb;13(2):209-21. doi: 10.1586/14779072.2015.1001368. Epub 2015 Jan 12. PMID 25578090
- [Result] Omboni S, Campolo L, Panzeri E. Telehealth in chronic disease management and the role of the Internet-of-Medical-Things: the Tholomeus(R) experience. Expert Rev Med Devices. 2020 Jul;17(7):659-670. doi: 10.1080/17434440.2020.1782734. Epub 2020 Jun 30. PMID 32536214
- [Result] Omboni S, Panzeri E, Campolo L. E-Health in Hypertension Management: an Insight into the Current and Future Role of Blood Pressure Telemonitoring. Curr Hypertens Rep. 2020 Jun 6;22(6):42. doi: 10.1007/s11906-020-01056-y. PMID 32506273
- [Result] Omboni S, McManus RJ, Bosworth HB, Chappell LC, Green BB, Kario K, Logan AG, Magid DJ, Mckinstry B, Margolis KL, Parati G, Wakefield BJ. Evidence and Recommendations on the Use of Telemedicine for the Management of Arterial Hypertension: An International Expert Position Paper. Hypertension. 2020 Nov;76(5):1368-1383. doi: 10.1161/HYPERTENSIONAHA.120.15873. Epub 2020 Sep 14. PMID 32921195
- [Result] Omboni S, Ballatore T, Rizzi F, Tomassini F, Campolo L, Panzeri E. Feasibility of 24-h blood pressure telemonitoring in community pharmacies: the TEMPLAR project. J Hypertens. 2021 Oct 1;39(10):2075-2081. doi: 10.1097/HJH.0000000000002895. PMID 34102664
- [Result] Omboni S, Ballatore T, Rizzi F, Tomassini F, Panzeri E, Campolo L. Telehealth at scale can improve chronic disease management in the community during a pandemic: An experience at the time of COVID-19. PLoS One. 2021 Sep 29;16(9):e0258015. doi: 10.1371/journal.pone.0258015. eCollection 2021. PMID 34587198
- [Result] Omboni S, Ballatore T, Rizzi F, Tomassini F, Campolo L, Panzeri E, Lundwall K, Kahan T. 24-hour ambulatory blood pressure telemonitoring in patients at risk of atrial fibrillation: results from the TEMPLAR project. Hypertens Res. 2022 Sep;45(9):1486-1495. doi: 10.1038/s41440-022-00932-1. Epub 2022 May 18. PMID 35585169
- [Result] Omboni S, Ballatore T, Rizzi F, Tomassini F, Campolo L, Panzeri E. Age-related patterns of ambulatory blood pressure in a large cohort of individuals referred to Italian community pharmacies: results from the templar project. J Hypertens. 2023 Feb 1;41(2):336-343. doi: 10.1097/HJH.0000000000003337. Epub 2022 Nov 28. PMID 36453645
- [Result] Omboni S. Reply to 'Extreme dipping: is the nocturnal blood pressure fall modulated by age?'. J Hypertens. 2023 May 1;41(5):868-869. doi: 10.1097/HJH.0000000000003388. No abstract available. PMID 37017033
- [Result] Omboni S, Khan NA, Kunadian V, Olszanecka A, Schutte AE, Mihailidou AS. Sex Differences in Ambulatory Blood Pressure Levels and Subtypes in a Large Italian Community Cohort. Hypertension. 2023 Jul;80(7):1417-1426. doi: 10.1161/HYPERTENSIONAHA.122.20589. Epub 2023 May 12. PMID 37315119
- See also: The official website of the TEMPLAR project with updates on the status of the study and current findings. — http://www.templarnet.org
- See also: The certified web-based telemedicine platform used to collect the data for the TEMPLAR Project. — http://www.tholomeus.net